CLINICAL TRIAL: NCT04208243
Title: Creative Arts Therapy (CAT) in the Center for Cancer and Blood Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-1028.cc
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Results first posted 2022-06-10 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The subjects and/or parents will be tested with all instruments before the intervention, and approximately every 30 days for no less than 3 months and a max participation of 6 months. Treatment time points will be at least 30 days apart. For those subjects who are scheduled to come into clinic every 1-2 months for SOC appointments, study participation may take up to 6 months. This 6 month time period would allow for the completion of 4 time points of CAT. The testing will take place in an exam room after vital signs have been completed upon intake. The study staff will administer the questionnaires. The PedsQL includes a subject report (ages 5 and over) and a parent report. The Resilience Scale is a self-report and will be used for ages 12 and over. The Faces Scale will use parent report for ages less than 5 and self-report for ages 5 and over. For consistency, the posture measure will be completed by study staff after training with the manual included with the inclinometer tool.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncology Patient (Experimental): Any Oncology patient in the CCBD who has not previously received more than two sessions of CAT in the outpatient unit and who will be receiving approximately weekly infusions of at least one hour in the infusion center will be identified by a research assistant.
  Interventions: Behavioral: Creative Arts Therapy

INTERVENTIONS:
Behavioral: Creative Arts Therapy — The intervention will consist of approximately weekly CAT in the infusion center during cancer therapy. The interventionist is a Master's prepared, licensed dance/movement therapist who is experienced in music and art therapies as well. The CAT includes dance/movement such as playing with a parachute, simple yoga breathing and postures, and work with physioballs. The music includes singing, listening to music, and playing instruments. The art consists of drawing, finger painting, working with clay. The CAT may occur in individual sessions in private infusion rooms, or in groups in the middle of the infusion center. The CAT is not only a distraction, but also a therapeutic process addressing the stressors of cancer and its treatment. The "dose" of CAT will be recorded (number and type of sessions) and will be factored into the analysis.

SUMMARY:
The purpose of the study is to evaluate the effectiveness of Creative Arts Therapy (CAT) on pediatric patients undergoing chemotherapy in the Infusion Center at Children's Hospital Colorado Center for Cancer and Blood Disorders. Findings from a previous pilot study support the hypothesis that CAT may improve quality of life (QOL), resiliency, physical posture, and emotional response to pain of pediatric oncology patients undergoing chemotherapy.

DETAILED DESCRIPTION:
A repeated measures design will be used with each patient serving as his/her own control. The subjects and/or parents will be tested with all instruments before the intervention, and approximately every 30 days for no less than 3 months and a maximum participation of 6 months. Treatment time points will be at least 30 days apart. Because some subjects are not scheduled to come into the clinic every 30 days for SOC appointments, they are unable to complete 3 sessions of CAT in a 3 month time period. For those subjects who are scheduled to come into clinic every 1-2 months for SOC appointments, study participation may take up to 6 months. This 6 month time period would allow for the completion of 4 different time points of CAT.

The testing will take place in an exam room after vital signs have been completed upon intake to the clinic. The trained research assistant, trained RN, or PI will administer the questionnaires. The PedsQL includes a subject report (ages 5 and over) and a parent report. The Resilience Scale is a self-report and will be used for ages 12 and over. The Faces Scale will use parent report for ages less than 5 and self-report for ages 5 and over. In order to confirm consistency, the posture measure will be completed by the PI (nurse practitioner) or registered nurse on the study after training with the manual included with the inclinometer tool.

ELIGIBILITY:
Inclusion Criteria:

* Center for Cancer and Blood Disorders (CCBD) patient with Oncology or Neuro-oncology diagnosis
* No more than 2 previous sessions of CAT as an outpatient in the CCBD
* English speaking
* Receiving outpatient chemotherapy, biotherapy, or transfusions in the infusion center approximately weekly for at least 3 months.
* Ages 3 to 18 years

Exclusion Criteria:

* Hematology or other patients in the infusion center
* Patients who have previously received more than 2 sessions of CAT in the infusion center
* Non-English speaking patients

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2010-09-29 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2023-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oncology Patient
Started | 83
Completed | 83
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oncology Patient
Number analyzed (Participants) | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 83
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 7.8 [3 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 79
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 83

OUTCOME MEASURES:

1. Primary Outcome: PedsQL 3.0 Cancer Module Scale
Description: The PedsQL 3.0 Cancer Module evolved from the PedsQL 4.0 Generic Core Scale. The instrument employs a Parent-Proxy Report for ages 2-18 years & a companion Child Self-Report for children 5 years and up. The Cancer Module is a 27-item instrument assessing 8 subscales (pain & hurt, nausea, procedural anxiety, treatment anxiety, worry, cognitive problems, perceived physical appearance, & communication). The PedsQL has been shown to be the most responsive to change when compared with other measures of QOL used with children undergoing chemotherapy. Reliability, assessed by internal consistency, yielded coefficient alphas ranging from .80-.90 across total & individual scales and are, thus, appropriate for group comparisons in this study. It is easily completed by parents in10 minutes and reverse-scored and linearly-transformed in five minutes. This tool uses a 0-100 score value system. The higher the score, the better the outcome. The subscales are summed to compute the total score.
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oncology Patient
Number analyzed (Participants) | 83
score on a scale | 71.59 (16.14)

2. Primary Outcome: The Resilience Scale (RS)
Description: The RS-14 is a 14-item scale using a 7-point rating (1-7). Higher scores mean superior levels of resilience tendencies, and each of the 14 items on the scale was summed to obtain a total score, so the theoretical full range is from 14 to 98. The construct of resilience is measured by two factors: personal competence and acceptance of self and life. Wagnild and Young have completed psychometric testing that established internal consistency reliability and concurrent validity. Many studies have validated that the scale may be used with samples of any age or ethnic background, but it is written at a 6th grade level. The authors who developed the tool are currently using it in adolescents. Given that it is expected that half the population of this study will be teenagers, this tool will be used with subjects ages 12 and over to obtain initial data on CAT's effect on resilience.
Time Frame: 7 months
Population: This scale is utilized only for patients 12 and older.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oncology Patient
Number analyzed (Participants) | 19
score on a scale | 82.86 (8.68)

3. Primary Outcome: McGrath Faces Scale
Description: The Faces Scale has been used for evaluating emotional responses to pain on children 3-17 years old. It is a one page form with nine faces in order of happy to upset. Numerical values are given to each face as determined by childrens' perspectives for an affective value by asking 200 children to directly scale the feelings depicted by the faces. The scale has been integrated as a routine measure for management of acute, recurrent, and chronic pain. For children under 3 years old, parents are asked to complete the Faces Scale. Although this scale has been used for emotional response to pain, it is felt to be an appropriate measure for the emotional response to the discomfort and anxiety in the infusion room. The scale has 9 faces scored from 1-9. The higher the number, the worse the pain. The scores are not summed or averaged, this tool has only 1 score with the range of 1 to 9. 1 is most positive emotional response and 9 is most negative emotional response.
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oncology Patient
Number analyzed (Participants) | 83
score on a scale | 2.89 (1.79)

4. Primary Outcome: Postural Measurement by Inclinometer
Description: Thoracic kyphosis will be measured using 2 gravity dependent inclinometers (Isomed Inc.). Spinal processes will be determined by palpation by a registered nurse or pediatric nurse practitioner. The feet of the inclinometers will be placed over the spinal processes thought to be at T1, T2 and T12, L1. The measurements will be taken in relaxed standing and measured 3 times in succession with the average of the 3 measures as the final value. Clinical assessment of the thoracic kyphosis angle is considered essential in postural examination, but can be time consuming when measured radiographically. The test-re-test reliability established excellent intra-rater reliability. Although validity of this measure is less studied, the measurement is thought to provide guidance of how much change of the kyphoscoliosis angle is a real consequence of intervention over time. Higher poster angle (from inclinometer) equals improved posture.
Time Frame: 7 months
Population: Participants were provided the option to decline the posture measure if the did not feel well enough to participate.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Oncology Patient
Number analyzed (Participants) | 68
degrees | 25.47 (9.22)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Oncology Patient
All-Cause Mortality (participants affected / at risk) | 0/83
Serious Adverse Events (participants affected / at risk) | 0/83
Other Adverse Events (participants affected / at risk) | 0/83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT04208243/Prot_SAP_ICF_000.pdf